CLINICAL TRIAL: NCT03826498
Title: Efficiency Evaluation of Allogenic Umbilical Cord Blood Mononuclear Cells (UCB-MNC) Transfusion in Patients With Autism
Brief Title: Allogenic Cord Blood Transfusion in Patients With Cerebral Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Responsible Party: Principal Investigator, Volchkov Stanislav, Deputy director, Quality assurance director, State-Financed Health Facility "Samara Regional Medical Center Dinasty"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12102017
Record Dates: First submitted 2019-01-22; First posted 2019-02-01 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; CP; Cord Blood; Stem cells
MeSH Terms: conditions — Cerebral Palsy | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CP CB-MNC injection (Experimental): CP CB-MNC injection from different donors and standard therapy.
  Interventions: Biological: CP CB-MNC injection; Other: Standard therapy
- Standard therapy (Other): Patients with standard therapy as control group
  Interventions: Other: Standard therapy

INTERVENTIONS:
Biological: CP CB-MNC injection — CB-MNC injection from different donors. One dose consist 20-50 mil MNC/kg.The protocol include 3 injection at monthly intervals.
  Arms: CP CB-MNC injection
Other: Standard therapy — The standard therapy can include drugs, special psychology training etc.

SUMMARY:
Cerebral palsy is a disorder of movement and posture resulted from a non-progressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability.

Many experimental animal studies have revealed that umbilical cord blood is useful to repair neurological injury in brain.

On the basis of many experimental studies, umbilical cord blood is suggested as a potential therapy for cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neurodevelopmental conditions with abnormal movement and posture resulted from a non-progressive cerebral disturbance. It is the most common cause of motor disability in childhood. Most therapies are palliative rather than restorative. Umbilical cord blood (UCB) may be used as restorative approach for children with CP.

Many experimental animal studies have revealed that UCB is beneficial to improve and repair neurological injuries, this effect achieved due to immune regulation and angiogenesis as well as the neuroprotective effect.

Based on animal studies and some clinical trials, UCB is suggested as a potential therapy for children with CP.

This study is prospective, non randomized (open label) with control group.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed diagnosis: Cerebral Palsy.

Exclusion Criteria:

* the presence of the following diseases in history: heart failure in the stage of decompensation, stroke in history less than 1 year ago, blood diseases;
* decompensation of chronic and endocrinological diseases;
* acute respiratory viral and bacterial infections, period less than 1 month after the acute phase.
* HIV infection, hepatitis B and C.
* oncological diseases, chemotherapy in the anamnesis;
* tuberculosis.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2024-01-26 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-serious and serious adverse events | 6 month
  Safety assessment such as adverse events will be registered. Adverse events will be monitored during all trial.
Changes in Standardized Gross Motor Function 66 (GMFM-66) Score for all child. | 1, 3, 6 month
  GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function). We reported changes of GMFM between each assessment time points. Categories of outcome table are baseline and values of just subtracting the latter raw scores from the former ones. This test will be acquired for all child.
Changes in Cognitive Neurodevelopmental Outcome for child before 3yrs | 1, 3, 6 month
  Bayley Scale of Infant Development-II (K-BSID-II) Mental Scales (higher value means better mental function: 0 - worst, 178 - best). We reported changes of BSID-II Mental Scale raw score between each assessment time points. Categories of outcome data are values of subtracting the latter scores from the former ones.This test will be acquired for child before 3yrs.
Changes in The Infant Toddler Quality of Life Questionnaire for child above 3yrs. | 1, 3, 6 month
  ITQOL - the 47-item short-form (ITQOL-SF47) developed for use in infants and toddlers from 2-months-to-5 years of age. Form scores physical, mental and social well being/ For each concept, item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health). Changes in completed questionnaire will be assessed. This test will be acquired for child above 3yrs.
Changes in Ashworth scale score for all child. | 1, 3, 6 month
  The Ashworth scale (AS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity scoring, where:
  0 No increase in tone;
  1. Slight increase in tone giving catch when the limb is moved in flexion and extension;
  2. More marked increase in tone, but limb is easily flexed;
  3. Considerable increases in tone, passive movement difficult;
  4. Limb rigid in flexion or extension. This test will be acquired for child above 3yrs.

SECONDARY OUTCOMES:
Number of Participants with Chimerism (longevity) of infused cell | 6 month
  Chimerism study to detect the longevity of infused donor cells and predict effectiveness of treatment. This study measure DNA of donor cells will in patients blood at the end of protocol. Absence of donor DNA suggest no chimerism.

CONTACTS AND LOCATIONS:
Overall Officials: STANISLAV VOLCHKOV, MD, PhD, Principal Investigator — Medical Centre Dinasty
Locations (1):
- Medical Centre Dinasty, Samara, Russia